CLINICAL TRIAL: NCT01014910
Title: Intermittent Versus Continuous Pulse Oximetry Monitoring of Infants Admitted for Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Baylor University (Other); Lifespan (Other); University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMTT# 4151-09
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Bronchiolitis; Hypoxia
Keywords: Bronchiolitis; Hypoxia; Pulse; Oximetry; Hospitalized
MeSH Terms: conditions — Bronchiolitis; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous pulse oximetry monitoring (Active Comparator): Patients will receive continuous pulse oximetry monitoring throughout their hospital stay regardless of their need for supplemental oxygen.
  Interventions: Other: Continuous pulse oximetry monitoring
- Intermittent pulse oximetry monitoring (Active Comparator): Patients will receive pulse oximetry monitoring during vital signs checks (every 4 hours) and as indicated clinically when not on supplemental oxygen. When patients require supplemental oxygen they will be continuously monitored by pulse oximetry until their oxygen requirement has resolved.
  Interventions: Device: Intermittent pulse oximetry monitoring

INTERVENTIONS:
Other: Continuous pulse oximetry monitoring — Placement of a pulse oximeter to monitor oxygenation status. This is usually placed on a toe, finger, or ear lobe and held in place with adhesive tape. Patients will receive continuous pulse oximetry monitoring throughout their hospital stay regardless of their need for supplemental oxygen.
  Other Names: Continuous pulse ox
  Arms: Continuous pulse oximetry monitoring
Device: Intermittent pulse oximetry monitoring — Placement of a pulse oximeter to monitor oxygenation status. This is usually placed on a toe, finger, or ear lobe and held in place with adhesive tape. Patients will receive pulse oximetry monitoring during vital signs checks (every 4 hours) and as indicated clinically when not on supplemental oxygen. When patients require supplemental oxygen they will be continuously monitored by pulse oximetry until their oxygen requirement has resolved.
  Other Names: Intermittent pulse ox
  Arms: Intermittent pulse oximetry monitoring

SUMMARY:
Bronchiolitis is a lower respiratory tract infection (LRTI) syndrome cause by different types of viruses and occurs in young children. Although bronchiolitis is a widespread and fairly common illness in children, pediatricians vary significantly in how it is treated. This includes how children are monitored for their oxygen status when not receiving supplemental oxygen. Studies suggest that continuous pulse oximetry measurement of children admitted to the hospital with bronchiolitis regardless of use of supplemental oxygen prolongs their hospital stay. This increases the cost of care for these patients and increases their risk of hospital-associated complications.

This study is a randomized trial of continuous pulse oximeter use in patients admitted with bronchiolitis versus transitioning patients not requiring oxygen to intermittent pulse oximetry monitoring. The investigators hypothesize that this will decrease length of stay as well as associated costs of care and number of medical interventions performed in the hospital.

DETAILED DESCRIPTION:
Background: Bronchiolitis is a lower respiratory tract infection (LRTI) syndrome caused by different viruses. It is the most common LRTI in children under 24 months old, accounting for approximately 90,000 hospitalizations annually and costing over $700 million in children under 12 months. Health care providers vary in diagnosis and management, however. In 2006 the American Academy of Pediatrics (AAP) released guidelines for bronchiolitis management in an effort to standardize clinical practice. Part of these guidelines recommends patients admitted to the hospital receive supplemental oxygen if they are persistently hypoxic, which is defined as pulse oximeter readings persistently below 90%. However, this recommendation is based on expert opinion.

Research has previously shown healthy infants routinely experience brief episodes of decreased oxygen levels while sleeping without significant health effects. Other studies demonstrate no relationship between short intervals of transient or mildly decreased oxygen levels and long-term mental or developmental delays. Furthermore, children with bronchiolitis remain hospitalized longer without any appreciable improvement in the course or outcome of their illness when continuously monitored for oxygen level.

Widespread pulse oximeter use has increased hospitalization rates over 250%, and close monitoring increases length of stay for children who otherwise could be discharged home. The 2006 guidelines discourage continuous pulse oximetry monitoring in children not requiring supplemental oxygen, but health care providers routinely ignore this recommendation. No studies have assessed the impact of more strictly adhering to the practices recommended by the AAP.

Research Procedures: This is a randomized control study and is a multi-site collaboration with University of Missouri Children's Hospital in Columbia, Missouri. Children admitted to the study sites with bronchiolitis will be batch randomized (i.e. randomized separately at each site) to undergo either continuous pulse oximetry monitoring throughout the entire hospitalization or receive intermittent monitoring when not on supplemental oxygen. Patients will additionally receive all care standard to the management of their illness. Of note, the proposed intervention is the recommended standard of care for oxygen monitoring compared to the general practice used at both study sites. Researchers will then review charts after discharge for length of stay, number of medical interventions performed, diagnostic testing completed, and treatments provided. Cost of stay for patients in each group will be estimated and compared as well. Patients will be involved in the study for their entire admission.

ELIGIBILITY:
Inclusion Criteria:

* Children less than or equal to 24 months old with a history of term delivery (gestational age ≥37 weeks) admitted with a presumptive diagnosis of bronchiolitis
* Bronchiolitis will be defined as an episode of wheezing or increased work of breathing associated with signs of an upper respiratory tract infection experienced by a patient
* Enrollment within 24 hours of admission

Exclusion Criteria:

* History of severe cardiac or pulmonary illness, including but not limited to bronchopulmonary dysplasia, chronic lung disease, asthma/reactive airway disease, congenital heart disease, heart failure, and cardiothoracic surgery
* History of home albuterol use for asthma or reactive airway disease
* History of use of bronchodilator with successful patient response to the medication
* Use of corticosteroids within the past two weeks up to day of admission
* Use of antibiotics after admission for suspected pneumonia or similar pulmonary disease
* History of premature birth (<37 weeks gestation)
* History of receiving palivizumab (anti-RSV antibody)
* Diagnosis of chronic immune deficiency, hematologic dyscrasia, or cancer
* Chronic treatment with immunosuppressants
* Parents/guardians unable to give informed consent in English
* Need for PICU transfer at any point during illness
* Transfer from an outside institution where patient was hospitalized for ≥12 hours
* Previous enrollment in this study
* Pediatric attending refuses to comply with study protocol

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2009-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Koster, MD, Principal Investigator — Hasbro Children's Hospital; Russell J McCulloh, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Vanessa Hill, MD, Principal Investigator — Christus Santa Rosa Children's Hospital
Locations (4):
- United States (4):
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Christus Santa Rosa Children's Hospital, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
IRB approval at participating institutions does not provide an avenue for sharing study data after study completion.

REFERENCES:
- [Background] Shay DK, Holman RC, Roosevelt GE, Clarke MJ, Anderson LJ. Bronchiolitis-associated mortality and estimates of respiratory syncytial virus-associated deaths among US children, 1979-1997. J Infect Dis. 2001 Jan 1;183(1):16-22. doi: 10.1086/317655. Epub 2000 Nov 10. PMID 11076709
- [Background] Willson DF, Horn SD, Hendley JO, Smout R, Gassaway J. Effect of practice variation on resource utilization in infants hospitalized for viral lower respiratory illness. Pediatrics. 2001 Oct;108(4):851-5. doi: 10.1542/peds.108.4.851. PMID 11581435
- [Background] Bass JL, Corwin M, Gozal D, Moore C, Nishida H, Parker S, Schonwald A, Wilker RE, Stehle S, Kinane TB. The effect of chronic or intermittent hypoxia on cognition in childhood: a review of the evidence. Pediatrics. 2004 Sep;114(3):805-16. doi: 10.1542/peds.2004-0227. PMID 15342857
- [Background] Hunt CE, Corwin MJ, Lister G, Weese-Mayer DE, Neuman MR, Tinsley L, Baird TM, Keens TG, Cabral HJ. Longitudinal assessment of hemoglobin oxygen saturation in healthy infants during the first 6 months of age. Collaborative Home Infant Monitoring Evaluation (CHIME) Study Group. J Pediatr. 1999 Nov;135(5):580-6. doi: 10.1016/s0022-3476(99)70056-9. PMID 10547246
- [Background] Bergman AB. Pulse oximetry: good technology misapplied. Arch Pediatr Adolesc Med. 2004 Jun;158(6):594-5. doi: 10.1001/archpedi.158.6.594. No abstract available. PMID 15184226
- [Background] Unger S, Cunningham S. Effect of oxygen supplementation on length of stay for infants hospitalized with acute viral bronchiolitis. Pediatrics. 2008 Mar;121(3):470-5. doi: 10.1542/peds.2007-1135. PMID 18310194
- [Background] Luo Z, Fu Z, Liu E, Xu X, Fu X, Peng D, Liu Y, Li S, Zeng F, Yang X. Nebulized hypertonic saline treatment in hospitalized children with moderate to severe viral bronchiolitis. Clin Microbiol Infect. 2011 Dec;17(12):1829-33. doi: 10.1111/j.1469-0691.2010.03304.x. Epub 2010 Jul 15. PMID 20636429
- [Background] Ralston S, Hill V, Martinez M. Nebulized hypertonic saline without adjunctive bronchodilators for children with bronchiolitis. Pediatrics. 2010 Sep;126(3):e520-5. doi: 10.1542/peds.2009-3105. Epub 2010 Aug 16. PMID 20713480
- [Derived] McCulloh R, Koster M, Ralston S, Johnson M, Hill V, Koehn K, Weddle G, Alverson B. Use of Intermittent vs Continuous Pulse Oximetry for Nonhypoxemic Infants and Young Children Hospitalized for Bronchiolitis: A Randomized Clinical Trial. JAMA Pediatr. 2015 Oct;169(10):898-904. doi: 10.1001/jamapediatrics.2015.1746. PMID 26322819

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from October 2009 to April 2014. Only 1 study site used an institutional clinical practice guideline during the study. Respiratory-distress scoring systems for hospitalized patients were not standardized across sites. All sites used an oxygen saturation level of 90% or higher in room air as a criterion for hospital discharge.
Pre-assignment Details: Participants were sequentially randomized at each site in strict chronological order of hospital admission each day. Screening of participants was performed on weekdays during normal business hours. only. Parents/guardians were blinded to allocation assignment until informed consent was obtained; study personnel and outcome assessors were not.
Period: Overall Study
Arm/Group | Continuous Pulse Oximetry Monitoring | Intermittent Pulse Oximetry Monitoring
Started | 80 | 81
Completed | 80 | 79
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Pulse Oximetry Monitoring | Intermittent Pulse Oximetry Monitoring | Total
Number analyzed (Participants) | 80 | 81 | 161
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 0.22 [0.13 to 0.44] | 0.30 [0.15 to 0.64] | 0.25 [0.13 to 0.52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 32 | 73
  Male | 39 | 49 | 88
Region of Enrollment [Number; unit: participants]
  United States | 80 | 81 | 161
Presence of rhonorrhea [Number; unit: participants] | 77 | 77 | 154
Decreased oral intake [Number; unit: participants] | 51 | 54 | 105
Vomiting [Number; unit: participants] | 32 | 40 | 72
Diarrhea [Number; unit: participants] | 14 | 14 | 28
Rash [Number; unit: participants] | 6 | 14 | 20
Irritability [Number; unit: participants] | 29 | 27 | 56
Lethargy [Number; unit: participants] | 12 | 11 | 23
Seizure [Number; unit: participants] | 0 | 0 | 0
History of tobacco exposure [Number; unit: participants] | 17 | 22 | 39
Family history of asthma/reactive airway disease [Number; unit: participants] | 30 | 45 | 75
Day-care exposure [Number; unit: participants] — Includes patients with a sibling in daycare
  participants | 8 | 15 | 23
Receipt of bronchodilators prior to admission [Number; unit: participants] | 58 | 63 | 121
Receipt of antibiotics prior to admission [Number; unit: participants] | 10 | 21 | 31
Receipt of oral corticosteroids before admission [Number; unit: participants] | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay in the Hospital
Time Frame: Summarized from admission to hospital discharge
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Continuous Pulse Oximetry Monitoring | Intermittent Pulse Oximetry Monitoring
Number analyzed (Participants) | 80 | 81
hours | 38.7 [23.6 to 64.7] | 39.5 [24.3 to 59.5]
Statistical Analysis 1: Comparison: Continuous Pulse Oximetry Monitoring vs Intermittent Pulse Oximetry Monitoring; Differences in LOS were compared between study arms using the Mann-Whitney U-test and the Kaplan-Meier method. Statistical analyses were performed using Stata version 13.1 for Windows (StataCorp). All patients enrolled in the study, including those who subsequently had consent for the intervention withdrawn, were included for analysis (intention to treat); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — Based on a previously-identified mean LOS of 65.3 hours, we estimated we would need to enroll 80 patients in each study arm to provide adequate sample size to detect a difference in mean LOS of 18 hours with 80% power and alpha=0.05; Sample size calculations were performed using Power and Sample Size Calculator, version 3.0 (by developers William D. Dupont and Walton D. Plummer Jr)

2. Secondary Outcome: Clinical Deterioration Necessitating Transfer to Higher Level of Care
Time Frame: Summarized from admission to hospital discharge
Measure: Number; unit: participants
Arm/Group | Continuous Pulse Oximetry Monitoring | Intermittent Pulse Oximetry Monitoring
Number analyzed (Participants) | 80 | 81
participants | 4 | 4
Statistical Analysis 1: Comparison: Continuous Pulse Oximetry Monitoring vs Intermittent Pulse Oximetry Monitoring; The proportion of patients transferred to the intensive care unit in each study arm was compared between study arms using the Pearson χ2 test. All patients enrolled in the study, including those who subsequently had consent for the intervention withdrawn, were included for analysis (intention to treat); Test type: Superiority or Other; p = 0.05, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected for the period of the patient's hospital stay as well as documentation of any hospital readmissions within 14 days of discharge from the hospital. No contact with patient families was made after hospital discharge.
Arm/Group | Continuous Pulse Oximetry Monitoring | Intermittent Pulse Oximetry Monitoring
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/81
Other Adverse Events (participants affected / at risk) | 0/80 | 0/81

LIMITATIONS AND CAVEATS:
Our study was not designed or powered to detect differences in ICU transfers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No